CLINICAL TRIAL: NCT03927885
Title: Open Labeled Placebo for Treatment of Cancer Related Fatigue in Patients With Advanced Cancer
Brief Title: Open Labeled Placebo in Reducing Cancer Related Fatigue in Patients With Advanced Cancer
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0526; NCI-2019-01027 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0526 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Advanced Malignant Solid Neoplasm; Metastatic Malignant Solid Neoplasm; Recurrent Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (open labeled placebo) (Experimental): Patients receive open labeled placebo PO BID for 4 weeks in the absence of disease progression.
  Interventions: Other: Placebo Administration; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (waiting list, open labeled placebo) (Active Comparator): Patients are assigned to a waiting list during week 1. Beginning in week 2, patients receive open labeled placebo PO BID for 3 weeks in the absence of disease progression.
  Interventions: Other: Placebo Administration; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Waiting List

INTERVENTIONS:
Other: Placebo Administration — Given open labeled placebo PO
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: Waiting List — Assigned to a waiting list
  Other Names: Waitlist
  Arms: Arm II (waiting list, open labeled placebo)

SUMMARY:
This phase II/III trial studies an open labeled placebo to see how well it works compared with waitlist control in reducing cancer related fatigue in patients with cancer that has spread to other places in the body. A placebo is not a drug and is not designed to treat any disease or illness. Recent studies have found that cancer related fatigue symptoms in cancer survivors are improved with open labeled placebo (that is, patients know they are taking a placebo). It is not yet known how well an open labeled placebo works when compared with waitlist control in reducing cancer related fatigue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the effects of open labeled placebo one tablet twice a day (OLP) compared to waitlist control (WLC) for reducing cancer-related fatigue (CRF) as measured by the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) subscale in fatigued advanced cancer patients at the end of one week.

SECONDARY OBJECTIVES:

I. To determine the preliminary efficacy open labeled placebo (OLP) and WLC on various fatigue dimensions - (Multidimensional Fatigue Symptom Inventory, MFSI-SF), depression (The Center for Epidemiologic Studies - Depression [CES-D]), cancer symptoms (Edmonton Symptom Assessment System [ESAS]), function and strength (six minute walk test, and 30-sec chair stand test), Global Symptom Evaluation (GSE), and quality of life (Functional Assessment of Cancer Therapy - General [FACT-G]) in these advanced cancer patients.

II. To determine effects of OLP on fatigue symptom composite score (ESAS fatigue, pain and depression) at the end of 1st and 4th week.

III. To examine the adherence and safety for the OLP as treatment for cancer related fatigue.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive open labeled placebo orally (PO) twice daily (BID) for 4 weeks in the absence of disease progression.

ARM II: Patients are assigned to a waiting list during week 1. Beginning in week 2, patients receive open labeled placebo PO BID for 3 weeks in the absence of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a diagnosis of advanced cancer (metastatic or recurrent incurable solid tumors)
* Presence of fatigue of >= 4/10 on Edmonton Symptom Assessment System (ESAS) Fatigue item (0-10 severity scale)
* Patient should describe fatigue as being present for a minimum of 2 weeks prior to screening
* Uncontrolled pain; patient is on opioids for the treatment of cancer pain, he/she must have had no major dose change (> 25%) for at least 48 hours prior to study entry. Change in opioid dose after study entry is allowed
* Patient must be 18 years of age or older. The questionnaires used in this study have been validated only in the adult population
* Patient must be willing to engage in telephone follow up with research staff
* Patient must have telephone access to be contacted by the research staff
* Hemoglobin level of >= 8 g/dL. Patient may receive packed red blood cell (PRBC) transfusion so as to have hemoglobin level of >= 8 g/dL so at participate in the study

Exclusion Criteria:

* Surgery, or pain relieving procedures within 2 weeks of entry into the study or during the study period
* Patients with history of substance abuse (Cut down, Annoyed, Guilty, Eye opener [CAGE] >= 2+), cognitively impaired (MD Anderson Symptom [MDAS] > 7)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-03-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in cancer related fatigue | Baseline up to 1 week
  Will use t-tests to assess the mean changes and standard deviations from baseline to follow-up between the groups.

SECONDARY OUTCOMES:
Change in quality of life (QOL) | Baseline up to 4 weeks
  Will use t-tests to assess the mean changes and standard deviations from baseline to follow-up between the groups. The percentage of patients who report 'better' in each group will be reported. Will also compare the % of patients who report 'somewhat better' to "a great deal better" in each group and report the difference between groups (chi-square tests).
Change in function strength | Baseline up to 4 weeks
  Will use t-tests to assess the mean changes and standard deviations from baseline to follow-up between the groups. The percentage of patients who report 'better' in each group will be reported. Will also compare the % of patients who report 'somewhat better' to "a great deal better" in each group and report the difference between groups (chi-square tests).
Change in Global Symptom Evaluation (GSE) | Baseline up to 4 weeks
  Will use t-tests to assess the mean changes and standard deviations from baseline to follow-up between the groups. The percentage of patients who report 'better' in each group will be reported. Will also compare the % of patients who report 'somewhat better' to "a great deal better" in each group and report the difference between groups (chi-square tests).
Changes in cluster composite scores of sleep disturbance | Baseline up to 1 week
  The primary comparison will be using changes in cluster composite scores of sleep disturbance from baseline to end of week 1 between the placebo arm and waitlist control arm. Exploratory graphical analysis of the data will be done. If the assumptions of the t-test are violated, will use the Wilcoxon rank sum test.
Changes in cluster composite scores of fatigue | Baseline up to 1 week
  The primary comparison will be using changes in cluster composite scores of fatigue from baseline to end of week 1 between the placebo arm and waitlist control arm. Exploratory graphical analysis of the data will be done. If the assumptions of the t-test are violated, will use the Wilcoxon rank sum test.
Changes in cluster composite scores of pain | Baseline up to 1 week
  The primary comparison will be using changes in cluster composite scores of pain from baseline to end of week 1 between the placebo arm and waitlist control arm. Exploratory graphical analysis of the data will be done. If the assumptions of the t-test are violated, will use the Wilcoxon rank sum test.
Changes in cluster composite scores of depression | Baseline up to 1 week
  The primary comparison will be using changes in cluster composite scores of depression from baseline to end of week 1 between the placebo arm and waitlist control arm. Exploratory graphical analysis of the data will be done. If the assumptions of the t-test are violated, will use the Wilcoxon rank sum test.
Adherence | Up to 4 weeks
  Will use a chi-square to test the difference in adherence between each placebo group versus waitlist control group.
Incidence of adverse events | Up to 4 weeks
  Will calculate the chi-square statistic to test the difference in adverse events between placebo group versus waitlist control group.

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Yennu, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org